CLINICAL TRIAL: NCT01637441
Title: Randomized Study Comparing Laparoscopic Sacropexy and Vaginal Mesh Surgery in Cystocele Repair
Brief Title: Prosthetic Pelvic Organ Prolapse Repair
Acronym: PROSPERE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2011_24; 2011-A01282-39 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2012-07-06; First posted 2012-07-11 (Estimated); Last update posted 2015-11-04 (Estimated); Status verified 2015-11

CONDITIONS: Cystocele
Keywords: bladder prolapse (cystocele); Pelvic organ prolapse repair; coelioscopic; prosthetic surgery; vaginal approach; Randomized study; laparoscopic sacropexy; vaginal mesh surgery; Stage II; Clavien Dindo
MeSH Terms: conditions — Cystocele | interventions — Laparoscopy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- laparoscopic sacropexy (Experimental): under laparoscopic vision, the vesico-vaginal space is dissected until the level of the bladder neck. a synthetic non absorbable mesh is placed between the bladder and the vagina. the mesh is sutured to the vagina and the apex (vaginal apex or uterus) and anchored to the prevertebral ligament in front of the promontorium.
  Interventions: Procedure: laparoscopic sacropexy
- vaginal mesh (Experimental): after anterior sagittal colpotomy, the bladder is dissected under the fascia layer, and the paravesical fossa are entered. a synthetic non absorbable mesh is placed with 4 arms suspension (trans obturator or not). treatment of the apex is mandatory.
  Interventions: Procedure: vaginal mesh

INTERVENTIONS:
Procedure: laparoscopic sacropexy — under laparoscopic vision, the vesico-vaginal space is dissected until the level of the bladder neck. a synthetic non absorbable mesh is placed between the bladder and the vagina. the mesh is sutured to the vagina and the apex (vaginal apex or uterus) and anchored to the prevertebral ligament in front of the promontorium.
  Other Names: laparoscopic surgery
  Arms: laparoscopic sacropexy
Procedure: vaginal mesh — after anterior sagittal colpotomy, the bladder is dissected under the fascia layer, and the paravesical fossa are entered. a synthetic non absorbable mesh is placed with 4 arms suspension (trans obturator or not). treatment of the apex is mandatory.
  Other Names: medical vaginal device
  Arms: vaginal mesh

SUMMARY:
The cystocele is the most frequent clinical shape of the genital prolapse. It is a frequent pathology in woman which can impair quality of life and generates pelvic, urinary or sexual functional disorders.

It's considered that 8 % of women will be undergo surgery in this indication before the age of 80 years. Numerous surgical techniques have been described and we distinguish the interventions according to the route (vaginal or abdominal), and according to the use or not of synthetic mesh (non-absorbable) to increase the anatomical results.

DETAILED DESCRIPTION:
This is a multicenter, randomized, comparative, 2-parallel-arm study in patients with pelvic organ prolapse (cystocele) Approximately 260 patients aged from 45 to 75 years will be allocated to have laparoscopic sacropexy or vaginal mesh surgery.

ELIGIBILITY:
Inclusion Criteria:

* Cystocele superior or equal to stage II of the international classification POP-Q, isolated or associated with other elements of prolapse.
* Patient must have provided written informed consent form prior to enrolment
* Patient must be insured

Exclusion Criteria:

* Previous of surgery for prolapse
* Unfavourable conditions to one or other of the 2 evaluated procedure
* Pelvic malignancy in the course of evolution
* Contraindication to the use of mesh
* Women not reading French
* Patients haven't have a social insurance
* Pregnancy or desire for future pregnancy
* To be under guardianship or deprived of liberty
* Simultaneous participation in another biomedical research

Ages: 45 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 262 (Actual)
Dates: Start 2012-09; Primary Completion 2015-07 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Morbidity (Dindo Classification) | 12 months
  Compare the morbidity of the sub-vesical synthetic mesh according to the route between laparoscopic sacropexy or vaginal in the symptomatic superior stage II cystoceles at 1 year follow-up.

SECONDARY OUTCOMES:
Specific complications | 12 months
  Comparison for the specific complications of sub-vesical mesh according to the route :
  * Symptomatic erosions, shrinkages, infections,
  * Serious Adverse event
Medium-term tolerance | 12 months
  Comparison of both techniques for the medium-term tolerance:
  * Sexual: sexual quality of life, de novo dyspareunia;
  * Urinary: urinary quality of life, urinary functional signs, urgenturia, leakage
  * Post-operative chronic pelvic pains
Clinical Efficiency | 12 months
  Comparison of both techniques for the medium-term (1 year follow-up)clinical efficiency:
  * rate of anatomical recurrences at one year,
  * functional Symptoms of prolapse, general quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Philippe LUCOT, MD, Principal Investigator — CHRU de LILLE
Locations (12):
- France (12):
  - Sébatien BLANC, Annecy
  - Hôpital Antoine Béclère, Clamart
  - CHU Estaing, Clermont-Ferrand
  - GCS Flandre Maritime, Grande-Synthe
  - CH La Rochelle Service de Gynécologie Obstétrique, La Rochelle
  - Hôpital BICETRE / Service de Gynécologie Obstétrique, Le Kremlin-Bicêtre
  - CHRU de Lille - Service de Gynécologie médico chirurgicale, Lille
  - CHU de Nîmes, Nîmes
  - Groupe Hospitalier Diaconesses Croix St-Simon, Paris
  - CHI Poissy-St-Germain / Service de gynécologie, Poissy
  - CHU de Poitiers, Poitiers
  - Hôpital de Hautepierre, Strasbourg